CLINICAL TRIAL: NCT01567852
Title: The Use of Ketamine Versus Methohexital for Electroconvulsive Therapy: A Cross-Over Comparative Study on Patient Recovery and Re-Orientation Time
Brief Title: Use of Ketamine vs Methohexital for Electroconvulsive Therapy (ECT) on Patient Recovery and Re-orientation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HRRC#: 11-236
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-06

CONDITIONS: Post-anesthesia Recovery; Orientation
Keywords: orientation; post-anesthesia recovery; electroconvulsive therapy
MeSH Terms: conditions — Orientation, Spatial | interventions — Ketamine; Methohexital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine First (Experimental): This arm will receive ketamine for induction first, followed by alternating treatments between methohexital and ketamine
  Interventions: Drug: Ketamine; Drug: Methohexital
- Methohexital First (Experimental): This arm will receive Methohexital first for induction, followed by alternating treatments between ketamine and methohexital.
  Interventions: Drug: Ketamine; Drug: Methohexital

INTERVENTIONS:
Drug: Ketamine — Ketamine (1.5mg/kg) will be given for induction, with room to titrate up to induction effect
Drug: Methohexital — Methohexital (1.5mg/kg) will be given for induction

SUMMARY:
When undergoing ECT treatments, patient recovery time and re-orientation time may be shorter using ketamine for induction than using methohexital.

DETAILED DESCRIPTION:
ECT treatments are done under general anesthesia, and the induction is commonly done with methohexital. We will study whether using ketamine as an induction agent will result in a faster recovery time and quicker re-orientation time compared to using methohexital.

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for ECT with a primary mood disorder (bipolar disorder, major depressive disorder) will be eligible to participate in this study. - Patients must have decisional capacity and must be able to consent for this study.

Exclusion Criteria:

* patients with a primary psychotic disorder (schizophrenia, schizoaffective disorder); patients designated as having an American Society of Anesthesiologist (ASA) Status of greater than 3;
* patients with a known allergic reactions to methohexital , ketamine and succinylcholine;
* patients with current or previous history of aneurysms, intracranial bleeds, or intracranial hypertension;
* patients with uncontrolled severe hypertension.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Yen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Then Methohexital (Alternating Each Trial): This arm will receive ketamine for induction first, followed by alternating treatments between methohexital and ketamine. Each induction is counted as one trial. Each trial is followed by a day of no treatment (2 days for weekends).
  Ketamine: Ketamine (1-1.5mg/kg) will be given for induction, with room to titrate up to induction effect
  Methohexital: Methohexital (1-1.5mg/kg) will be given for induction, with room to titrate up to induction effect
- Methohexital Then Ketamine (Alternating Each Trial): This arm will receive Methohexital first for induction, followed by alternating treatments between ketamine and methohexital. Each induction is one trial. Each trial is followed by one day of no treatment (2 days for weekends).
  Ketamine: Ketamine (1-1.5mg/kg) will be given for induction, with room to titrate up to induction effect
  Methohexital: Methohexital (1-1.5mg/kg) will be given for induction, with room to titrate up to induction effect
Period: Overall Study
Arm/Group | Ketamine Then Methohexital (Alternating Each Trial) | Methohexital Then Ketamine (Alternating Each Trial)
Started | 8 | 12
Completed | 4 | 5
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 3 | 6
Not completed — ECT discontinued | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ketamine First: This arm will receive ketamine for induction first, followed by alternating treatments between methohexital and ketamine
  Ketamine: Ketamine (1-1.5mg/kg) will be given for induction, with room to titrate up to induction effect
  Methohexital: Methohexital (1-1.5mg/kg) will be given for induction
- Methohexital First: This arm will receive Methohexital first for induction, followed by alternating treatments between ketamine and methohexital.
  Ketamine: Ketamine (1-1.5mg/kg) will be given for induction, with room to titrate up to induction effect
  Methohexital: Methohexital (1-1.5mg/kg) will be given for induction
- Total: Total of all reporting groups
Arm/Group | Ketamine First | Methohexital First | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.75 (13.46) | 54 (22.63) | 52.65 (17.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Re-orientation Time
Description: Patients will be scored based on 5 questions (name, age, year, day of week, location). Each patient will be scored prior to induction as to how many questions they score correctly. Patient is deemed re-oriented when they score the same as baseline after the treatment.
Time Frame: 1 hour
Population: Since this was a crossover study, all patients received both drugs, except for 2 patients who dropped out after receiving the first drug. For one of these patients the drug was ketamine, for the other the drug was methohexital. Number of total trials analyzed was 69, with 35 Ketamine trials and 34 Methohexital trials
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Ketamine Inductions: Patients receiving Ketamine inductions for ECT
- Methohexital Inductions: Patients receiving methohexital for inductions
Arm/Group | Ketamine Inductions | Methohexital Inductions
Number analyzed (Participants) | 19 | 19
minutes | 24.5 (1.6) | 19.5 (1.6)

2. Primary Outcome: Recovery Time
Description: Recovery was assessed using 5 criteria (blood pressure, voluntary movement, oxygen requirement, consciousness, respiratory effort). Each criteria was scored from 0-2, with a full score of 10. The patient is scored at baseline, and is deemed recovered when all criteria has reached baseline score again.
Time Frame: 1 hour
Population: Please see description from outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ketamine Inductions | Methohexital Inductions
Number analyzed (Participants) | 19 | 19
minutes | 28.6 (2.0) | 27.2 (1.7)

ADVERSE EVENTS:
Description: Due to the cross-over, the same participant experienced different adverse effects according to which medication they received for induction. Hence, the number of adverse events is reported per trial (each trial is one induction) instead of per participant. There was a total of 35 trials with ketamine, and 34 trials with methohexital.
Groups:
- Ketamine Inductions: Number of trials receiving ketamine inductions. Each trial is one induction.
- Methohexital Inductions: Number of trials receiving methohexital inductions. Each trial is one induction
Arm/Group | Ketamine Inductions | Methohexital Inductions
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 19/35 | 8/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine Inductions (N=35) | Methohexital Inductions (N=34)
Nausea (Gastrointestinal disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Dysphoria (Psychiatric disorders) | 4 | 0
Headache (General disorders) | 2 | 1
Anesthesia Awareness (General disorders) | 0 | 1
Dizziness (General disorders) | 3 | 2
Agitation (Psychiatric disorders) | 1 | 0
Lethargy (General disorders) | 2 | 2
Hallucination (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No